CLINICAL TRIAL: NCT04378608
Title: Efficacy of Ombitasvir With Paritaprevir/Ritonavir Plus Ribavirin on the Treatment naïve Patients With Chronic Hepatitis C Virus Genotype 4
Brief Title: Ombitasvir /Paritaprevir/Ritonavir Plus Ribavirin on HCV GT4
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qu2018
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C Virus Infection
Keywords: Ombitasvir; Paritaprevir; Ritonavir; Ribavirin; HCV; Genotype 4; Naïve; Egyptians
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; paritaprevir; ombitasvir

STUDY DESIGN:
Intervention Model Description: 100 Egyptian naive patients infected with HCV GT4 was allocated and administered orally OBV/PTV/r with RBV which given as oral tablets based on patient tolerability
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2 DAA (OBV/PTV/r) ± ribavirin (RBV) (Other): Administering Ombitasvir/Paritaprevir/Ritonavir/ tablets plus RBV tablets to HCV GT4 in the treatment of Egyptian naïve patients
  Interventions: Drug: OBV/PTV/r) ± ribavirin (RBV)

INTERVENTIONS:
Drug: OBV/PTV/r) ± ribavirin (RBV)
  Other Names: Paritaprevir (ABT-450) is inhibitor of the NS3-4A serine protease Ombitasvir (ABT 267) is an NS5A inhibitor

SUMMARY:
The objective of the investigators was to delineate the efficacy and safety of Ombitasvir, paritaprevir with ritonavir (OBV/PTV/r) plus ribavirin (RBV) on chronic HCV GT4 Egyptian naïve patients

DETAILED DESCRIPTION:
Direct-acting antivirals (DAAs) combination therapies from various mechanisms of action and families have been revolutionized the management landscape of chronic hepatitis C virus (HCV). Ombitasvir, paritaprevir with ritonavir (OBV/PTV/r) ± ribavirin (RBV) are approved to treat HCV genotype 4 (GT4) infection. Here, investigators' objective was to delineate the efficacy and safety of OBV/PTV/r plus RBV of HCV GT4 in the treatment of Egyptian naïve patients.

Between 5 January and 8 September 2017, a cohort of 100 Egyptian patients infected with HCV GT4 was allocated and administered orally OBV/PTV/r with RBV, for 12 weeks, which given as oral tablets based on patient tolerability. The primary endpoint of investigators' study was a sustained virological response (HCV RNA < 12 IU/mL) 12 weeks from the cessation of the treatment (SVR12).

ELIGIBILITY:
Inclusion Criteria:

Treatment-naïve patients with HCV GT4 with plasma HCV RNA level >10,000 IU/ml

Exclusion Criteria:

* Hepatitis of non-HCV cause
* Coinfection with other than HCV GT4
* Poorly controlled diabetics (HbA1C >8) patients
* a history of extra-hepatocellular malignancy in the last 5 years
* Major severe illness such as congestive heart failure, respiratory failure, evidence of hepatic decompensation.
* Laboratory and blood picture abnormalities such as anemia (hemoglobin concentration of 10 <g/dl) and thrombocytopenia (platelets <50,000 cells/mm3) and (serum albumin <2.8 g/dL, international normalized ratio (INR) of > 2.3, serum total bilirubin concentration of >3.0 mg/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) | 12 weeks after last dose
  SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than 12 IU/mL 12 weeks after the last dose of study drug.
adverse event (AE) | Screening up to 30 days after last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation observed after administering a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is an event that results in, death, participant hospitalization, life-threatening, significant disability/incapacity, or a congenital anomaly.

SECONDARY OUTCOMES:
Percentage of Participants With Post-treatment Relapse Within 12 Weeks Following End of Treatment | Up to 12 weeks after last dose
  Post-treatment relapse was defined as defined as confirmed HCV RNA > 12 IU/ml between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < 12 IU/ml at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdel-Gabbar, Ass. Prof, Principal Investigator — Biochemistry Dep., Faculty of Science, Beni-Suef University, P.O. Box 52621

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Moneim A, Aboud A, Abdel-Gabbar M, Zanaty M, Ramadan M. Retreatment Efficacy of Sofosbuvir/Ombitasvir/Paritaprevir/Ritonavir + Ribavirin for Hepatitis C Virus Genotype 4 Patients. Dig Dis Sci. 2018 May;63(5):1341-1347. doi: 10.1007/s10620-018-5005-8. Epub 2018 Mar 15. PMID 29546644
- See also: This link clarify the retreatment efficacy and safety of SOF with OBV/PTV/r + RBV, for chronic HCV GT4-experienced patients who failed treatment with DAA-based regimens — https://doi.org/10.1007/s10620-018-5005-8